CLINICAL TRIAL: NCT05577520
Title: Maxillary Sinus Augmentation Using Different Size Bovine Bone Particles: a Histomorfometric Comparison
Brief Title: Maxillary Sinus Augmentation Using Different Size Bovine Bone Particles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Salvador, Argentina (Other)
Responsible Party: Principal Investigator, Jorge Ernesto Aguilar, Director and Professor, Oral Implantology Program, Universidad del Salvador, Argentina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRDI 1801
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Maxillary Sinus Augmentation
Keywords: Sinus floor augmentation; Xenograft; Anorganic; Bovine bone; Histomorphometry
MeSH Terms: interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: Small particle group (SPG n=10): MSA using 250 to 1000 µm size ABBM particles (Osteodens®, Pharmatrix, Argentina) as bone substitute.
  Large particles group (LPG n=10): MSA using 1000 to 2000 µm size ABBM particles (Osteodens®, Pharmatrix, Argentina) as bone substitute.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small particle group (SPG) (Experimental): SPG (n=10): MSA using 250 to 1000 µm size ABBM particles (Osteodens®, Pharmatrix, Argentina) as bone substitute.
  Interventions: Procedure: Sinus floor augmentation
- Large particles group (LPG) (Experimental): LPG (n=10): MSA using 1000 to 2000 µm size ABBM particles (Osteodens®, Pharmatrix, Argentina) as bone substitute.
  Interventions: Procedure: Sinus floor augmentation

INTERVENTIONS:
Procedure: Sinus floor augmentation
  Other Names: Sinus floor lift; Sinus floor elevation

SUMMARY:
The decrease in maxillary alveolar ridge bone volume and sinus pneumatization are a challenge to implant-assisted prosthetic rehabilitation. Guided bone regeneration using bone substitutes is an adequate alternative for maxillary sinus augmentation. Objective: To histologically and histomorphometrically compare bone repair response to 250 to 1000 µm and 1000 to 2000 µm anorganic bovine bone mineral (ABBM) particles as bone substitute in maxillary sinus augmentation (MSA).

DETAILED DESCRIPTION:
Twenty patients were treated with SMA in two steps. They were randomly assigned to one of two groups (n=10): SPG (small particles group) and LPG (large particles group). Different size ABBM particles were implanted in their maxillary sinus, accordingly. A vertical bone core biopsy was obtained at the implant site using a punch trephine. The samples were processed for histological observation and measured histomorphometrically to determine the percentage onewly formed bone (%NB), bone substitute (%BS), bone marrow (%BM), and osseointegration (%OI). Results were statistically analyzed using Student's t test (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 21 years
* Patients missing teeth in the maxillary sinus region (uni- or bilaterally) with a residual subantral bone height ≤ 4 mm and an alveolar ridge width ≥ 6mm.
* Patients who had not undergone tooth extraction within 6 months prior to enrollment.

Exclusion Criteria:

* Patients with diabetes, blood discrasias, a history of head and neck chemotherapy/radiation therapy, acute sinusitis or a history of allergic sinusitis, chronic polypoid sinusitis, or sinus tumors, or a history of Caldwell-Luc surgery
* Women who were pregnant or of childbearing age
* Alcoholics and drug abusers
* Patients requiring MS treatment showing anatomical features of the MS that contraindicated the surgical treatment
* Patients who refused to sign the informed consent form

Patients with a history of chronic periodontitis were treated and then enrolled in the study. Patients who developed post-operative maxillary sinus infection or showed allergic reactions attributable to the grafting material were eliminated from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of newly formed bone (NB) | 10 month
  histomorphometric parameter was assessed in a standardized area
Percentage of bone substitute | 10 month
  histomorphometric parameter was assessed in a standardized area
Percentage of bone marrow | 10 month
  histomorphometric parameter was assessed in a standardized area
Percentage of osseointegration | 10 month
  histomorphometric parameter was assessed in a standardized area, defined as the percentage of graft particle-newly formed bone integration

CONTACTS AND LOCATIONS:
Overall Officials: jorge aguilar, Chair Prof., Principal Investigator — Salvador University /Argentine Dental Association (USAL/AOA); Sandra Renou, Assoc. Prof., Study Director — Buenos Aires University (Argentine); Alicia Labandeira, Chair Prof., Principal Investigator — Salvador University /Argentine Dental Association (USAL/AOA); Maria Piloni, Assoc. Prof., Principal Investigator — Buenos Aires University (Argentine)
Locations (1):
- Masters in Dental Implantology (MIO) program at the University of Salvador (USAL)-Argentine Dental Association, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Fabbro M, Testori T, Francetti L, Weinstein R. Systematic review of survival rates for implants placed in the grafted maxillary sinus. Int J Periodontics Restorative Dent. 2004 Dec;24(6):565-77. PMID 15626319
- [Result] Smiler DG, Johnson PW, Lozada JL, Misch C, Rosenlicht JL, Tatum OH Jr, Wagner JR. Sinus lift grafts and endosseous implants. Treatment of the atrophic posterior maxilla. Dent Clin North Am. 1992 Jan;36(1):151-86; discussion 187-8. PMID 1737600
- [Result] Wallace SS, Froum SJ. Effect of maxillary sinus augmentation on the survival of endosseous dental implants. A systematic review. Ann Periodontol. 2003 Dec;8(1):328-43. doi: 10.1902/annals.2003.8.1.328. PMID 14971260
- [Result] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Result] Cricchio G, Sennerby L, Lundgren S. Sinus bone formation and implant survival after sinus membrane elevation and implant placement: a 1- to 6-year follow-up study. Clin Oral Implants Res. 2011 Oct;22(10):1200-1212. doi: 10.1111/j.1600-0501.2010.02096.x. PMID 21906186
- [Result] Bornstein MM, Chappuis V, von Arx T, Buser D. Performance of dental implants after staged sinus floor elevation procedures: 5-year results of a prospective study in partially edentulous patients. Clin Oral Implants Res. 2008 Oct;19(10):1034-43. doi: 10.1111/j.1600-0501.2008.01573.x. PMID 18828820
- [Result] Boyne PJ, James RA. Grafting of the maxillary sinus floor with autogenous marrow and bone. J Oral Surg. 1980 Aug;38(8):613-6. No abstract available. PMID 6993637
- [Result] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Result] Pejrone G, Lorenzetti M, Mozzati M, Valente G, Schierano GM. Sinus floor augmentation with autogenous iliac bone block grafts: a histological and histomorphometrical report on the two-step surgical technique. Int J Oral Maxillofac Surg. 2002 Aug;31(4):383-8. doi: 10.1054/ijom.2002.0286. PMID 12361071
- [Result] van den Bergh JP, ten Bruggenkate CM, Krekeler G, Tuinzing DB. Sinusfloor elevation and grafting with autogenous iliac crest bone. Clin Oral Implants Res. 1998 Dec;9(6):429-35. doi: 10.1034/j.1600-0501.1996.090608.x. PMID 11429944
- [Result] Chackartchi T, Iezzi G, Goldstein M, Klinger A, Soskolne A, Piattelli A, Shapira L. Sinus floor augmentation using large (1-2 mm) or small (0.25-1 mm) bovine bone mineral particles: a prospective, intra-individual controlled clinical, micro-computerized tomography and histomorphometric study. Clin Oral Implants Res. 2011 May;22(5):473-80. doi: 10.1111/j.1600-0501.2010.02032.x. Epub 2010 Nov 19. PMID 21087317
- [Result] Pebé PJ, Ramos A, Beovide AV, Borgia G, Ravecca T. Ensayo clínico aleatorizado de elevación sinusal por abordaje lateral con hueso mineral bovino desproteinizado (hmbd) comparando dos tamaños de partículas: resultados clínicos e histológicos. Odontoestomatología. 2017;19:57-67.
- [Result] de Molon RS, Magalhaes-Tunes FS, Semedo CV, Furlan RG, de Souza LGL, de Souza Faloni AP, Marcantonio E Jr, Faeda RS. A randomized clinical trial evaluating maxillary sinus augmentation with different particle sizes of demineralized bovine bone mineral: histological and immunohistochemical analysis. Int J Oral Maxillofac Surg. 2019 Jun;48(6):810-823. doi: 10.1016/j.ijom.2018.09.003. Epub 2018 Nov 13. PMID 30442550
- [Result] Testori T, Wallace SS, Trisi P, Capelli M, Zuffetti F, Del Fabbro M. Effect of xenograft (ABBM) particle size on vital bone formation following maxillary sinus augmentation: a multicenter, randomized, controlled, clinical histomorphometric trial. Int J Periodontics Restorative Dent. 2013 Jul-Aug;33(4):467-75. doi: 10.11607/prd.1423. PMID 23820706